CLINICAL TRIAL: NCT03768362
Title: Comparison of Medial Rectus Resection and Plication in Exotropic Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamideh Sabbaghi, PhD student, Teacher Assistant, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13112
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Exotropia
MeSH Terms: conditions — Exotropia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Undergoing plication strabismus surgery (Experimental)
  Interventions: Procedure: Plication strabismus surgery
- Undergoing resection strabismus surgery (Active Comparator)
  Interventions: Procedure: Resection strabismus surgery

INTERVENTIONS:
Procedure: Plication strabismus surgery — The technique was the same as resection up to muscle suturing, in the next step, the sutures were passed through 2 scleral bites at 1 mm anterior to the muscle insertion, then the muscle was folded toward inside or outside by pulling and joining the sutures. At the end, conjunctiva was repaired by vicryl 8/0.
  Arms: Undergoing plication strabismus surgery
Procedure: Resection strabismus surgery — resection strabismus surgery
  Arms: Undergoing resection strabismus surgery

SUMMARY:
Purpose: To determine the surgical outcomes of the plication technique in comparison with the resection method on exotropic patients.

Methods: In this randomized clinical trial, a total of 52 exotropic patients (female, 51.9%) who are candidate for medial rectus strengthening will be randomly classified into plication (n=24) and resection (n=28) groups. The comprehensive visual and ocular examinations will be performed on all study subjects and they will be followed- up for three months postoperatively. Plication technique is the same as resection up to muscle suturing, in the next step, the sutures are passed through 2 scleral bites at 1 mm anterior to the muscle insertion, then the muscle was folded toward inside or outside by pulling and joining the sutures.

ELIGIBILITY:
Inclusion Criteria:

Patients with a residual exotropia and history of uni- or bilateral lateral rectus recession or recession and resection (R &R) and those exotropic patients who were going to have already recession and resection (R & R) operation due to unilateral constant exotropia will be considered as eligible cases to be included.

Exclusion Criteria:

Subjects with a history of prematurity, intellectual disability, lack of central fixation (nystagmus, eccentric fixation, retinopathy of prematurity) subjects with systemic or other ocular diseases, neurological disorders, uncooperative patients and participants with less than three-month postoperative follow-up will be excluded from this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 52 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Postoperative ocular deviation | three months
  Postoperative ocular deviation will be measured at a distance of 6 meters three months after the surgery.

IPD SHARING:
Plan to Share IPD: Undecided